CLINICAL TRIAL: NCT06207539
Title: Use Of Hyoscine as An Adjuvant Treatment on Shortening the Time of Abortion Induction in Second Trimester: Randomized Controlled Clinical Trial
Brief Title: Induction of Abortion in the Second Trimester
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Ain Shams Maternity Hospital (Other)
Responsible Party: Principal Investigator, Andrew Nader Sed, Doctor, Ain Shams Maternity Hospital
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Supportive Care
Other Study IDs: Abortion
Record Dates: First submitted 2024-01-05; First posted 2024-01-17 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2022-12

CONDITIONS: Abortion, Second Trimester

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Other): Intramuscular administration of 20 milligrams hyoscine N-butyl bromide under the generic name of buscopan ampoule produced by Sanofi company, plus misoprostol under the generic name of misotac tablets, each of wich is 200 micrograms produced by Sigma company, approximately 400 micrograms (2 tablets) given by a member of the study team according to FIGO guidelines for use of misoprostol 2019 and to have a halved dose to 200 micrograms if patient with history of one or two cesarean section.
  Misoprostol only will be repeated every 4 hours for maximum 5 doses.
  Interventions: Drug: hyoscine N-butyl bromide under the generic name of buscopan ampoule produced by Sanofi company; Drug: misoprostol under the generic name of misotac tablets
- Group 2 (Other): Administration of misoprostol under generic name of misotac tablets each one is 200 micrograms produced by Sigma company, about 400 micrograms (2 tablets) given by a member of the study team according to FIGO guidelines use of misoprostol 2019 and to have a halved dose if patient with history of one or two cesarean sections.
  Misoprostol only will be repeated every 4 hours for maximum 5 doses.
  Interventions: Drug: misoprostol under the generic name of misotac tablets

INTERVENTIONS:
Drug: hyoscine N-butyl bromide under the generic name of buscopan ampoule produced by Sanofi company — compare between the effects of misoprostol with hyoscine N-butyl bromide and misoprostol alone on shortening the time of abortion induction in the second trimester.
  Other Names: Buscopan ampules
  Arms: Group 1
Drug: misoprostol under the generic name of misotac tablets — compare between the effects of misoprostol with hyoscine N-butyl bromide and misoprostol alone on shortening the time of abortion induction in the second trimester.
  Other Names: Misotac tablets

SUMMARY:
To compare between the effects of misoprostol with hyoscine N-butyl bromide and misoprostol alone on shortening the time of abortion induction in the second trimester.

DETAILED DESCRIPTION:
The study will be conducted on 40 women who will undergo induction of abortion between 13-24 weeks with positive fetal pulsation. They will be randomly assigned to receive either only misoprostol 400 μg under the generic name of misotac tablets produced by Sigma company according to FIGO classification 2019 and a halved dose if the patient has a history of one or two cesarean sections, or misoprostol 400 μg plus intramuscular administration of hyoscine N-butyl bromide under the generic name of buscopan ampoule produced by Sanofi company.

ELIGIBILITY:
Inclusion Criteria:

1. Abortion between 13-24 weeks with positive fetal pulsation due to congenital fetal malformations, severe preeclampsia, and maternal life-threatening conditions.
2. Women have up to two cesarean sections.

Exclusion Criteria:

1. Abortion between 13-24 weeks with no fetal pulsation
2. Women who have had two or more caesarean sections.
3. Multiple pregnancies
4. Uterine anomalies, such as septate and didelphis uteri.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-03-30 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
Efficacy of hyoscine as an adjuvant treatment in second trimester abortion | Baseline
  Admission Abortion interval (duration from the admission up to initiation of abortion).

CONTACTS AND LOCATIONS:
Overall Officials: Rania G Anwar El-Skaan, Study Director — Lecturer of Obstetrics and Gynecology, Faculty of Medicine, Ain Shams University
Locations (1):
- Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Allen R, O'Brien BM. Uses of misoprostol in obstetrics and gynecology. Rev Obstet Gynecol. 2009 Summer;2(3):159-68. PMID 19826573
- [Background] Stephenson ML, Wing DA. A novel misoprostol delivery system for induction of labor: clinical utility and patient considerations. Drug Des Devel Ther. 2015 Apr 22;9:2321-7. doi: 10.2147/DDDT.S64227. eCollection 2015. PMID 25960635
- See also: Effect of hyoscine butylbromide on cervical dilation during labor Medicina Universitaria — https://www.elsevier.es/es-revista-medicina-universitaria-304-articulo-effect-hyoscine-butylbromide-on-cervical-S1665579615000022